CLINICAL TRIAL: NCT00085475
Title: Phase II Study of Glivec (Imatinib) in Locally Advanced and/or Metastatic Soft Tissue Sarcomas Expressing the t(17;22)(q22;q13) Translocation Resulting in a COL1A1/PDGF-beta Fusion Protein i.e. DermatoFibroSarcoma Protuberans (DFSP) and Giant Cell Fibroblastoma (GCF)
Brief Title: Imatinib Mesylate in Treating Patients With Locally Advanced or Metastatic Dermatofibrosarcoma Protuberans or Giant Cell Fibroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-62027; EORTC-62027; EUDRACT-2004-002538-20
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; adult fibrosarcoma; adult malignant fibrous histiocytoma
MeSH Terms: conditions — Sarcoma; Fibrosarcoma; Histiocytoma, Malignant Fibrous | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: imatinib mesylate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase II trial is studying how well imatinib mesylate works in treating patients with locally advanced or metastatic dermatofibrosarcoma protuberans or giant cell fibroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the therapeutic activity of imatinib mesylate in patients with locally advanced or metastatic dermatofibrosarcoma protuberans or giant cell fibroblastoma.
* Determine the progression-free rate at 14 weeks in patients treated with this drug.

Secondary

* Determine objective response rate, progression-free survival, and overall survival in patients treated with this drug.
* Determine the duration of response in patients treated with this drug.

OUTLINE: This is an open-label, non-randomized, multicenter study.

Patients receive oral imatinib mesylate twice daily for at least 14 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 14 weeks receive imatinib mesylate for 12 additional weeks. Patients with a partial or complete response at 14 weeks undergo surgical resection if possible. If surgical resection of all remaining tumor is not possible OR if complete resection is not achieved (section margins positive), patients continue to receive imatinib mesylate in the absence of disease progression

Patients are followed monthly for 6 months, every 3 months for 6 months, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed dermatofibrosarcoma protuberans or giant cell fibroblastoma

  * Locally advanced or metastatic disease
* Measurable disease
* Not amenable to surgery, radiotherapy, or combined modality therapy with curative intent
* Documented progressive disease within the past 3 months

  * Previously irradiated lesions must show disease progression
* Tumor expressing COL1A1/PDGF-beta by fluorescence in situ hybridization

  * Translocation t(17;22)(q22;q13)
* No prior chemotherapy OR previously treated with 1, and only 1, line of combination chemotherapy with ifosfamide and doxorubicin OR 2 lines of single-agent therapy OR relapsed within 6 months after adjuvant chemotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 mg/dL* NOTE: *Transfusion allowed

Hepatic

* SGOT or SGPT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if hepatic metastases are present)
* Bilirubin ≤ 1.5 times ULN
* No uncontrolled hepatic disease

Renal

* Creatinine ≤ 1.5 times ULN
* No uncontrolled renal disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* HIV negative
* No uncontrolled diabetes
* No active or uncontrolled infection
* No concurrent severe or uncontrolled medical disease
* No medical, psychological, familial, sociological, or geographical condition that would preclude study participation, compliance, or giving informed consent
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 28 days since prior biologic therapy
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)
* No concurrent anticancer biologic agents

Chemotherapy

* See Disease Characteristics
* More than 28 days since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 6 months since prior radiotherapy
* No concurrent radiotherapy

  * Concurrent palliative radiotherapy allowed provided radiotherapy will not be administered to a target lesion

Surgery

* Not specified

Other

* More than 28 days since prior investigational drugs
* No concurrent therapeutic anticoagulation therapy with warfarin

  * Concurrent low-molecular weight heparin or mini-dose warfarin for prophylaxis of central venous catheter thrombosis allowed
* No other concurrent anticancer agents
* No other concurrent investigational drugs
* No other concurrent cytostatic agents
* No other concurrent tyrosine kinase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-04; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Progression-free rate at 14 weeks

SECONDARY OUTCOMES:
Response rate as assessed by RECIST criteria
Progression-free survival
Overall survival
Duration of response
Toxicity as assessed by CTC 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Allan T. van Oosterom, MD, PhD, Study Chair — University Hospital, Gasthuisberg
Locations (7):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - U.Z. Gasthuisberg, Leuven
- France (2):
  - Institut Bergonie, Bordeaux
  - CHU de la Timone, Marseille
- Netherlands (2):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Leiden University Medical Center, Leiden
- Christie Hospital NHS Trust, Manchester, England, United Kingdom

REFERENCES:
- [Background] Rutkowski P, Van Glabbeke M, Rankin CJ, Ruka W, Rubin BP, Debiec-Rychter M, Lazar A, Gelderblom H, Sciot R, Lopez-Terrada D, Hohenberger P, van Oosterom AT, Schuetze SM; European Organisation for Research and Treatment of Cancer Soft Tissue/Bone Sarcoma Group; Southwest Oncology Group. Imatinib mesylate in advanced dermatofibrosarcoma protuberans: pooled analysis of two phase II clinical trials. J Clin Oncol. 2010 Apr 1;28(10):1772-9. doi: 10.1200/JCO.2009.25.7899. Epub 2010 Mar 1. PMID 20194851